CLINICAL TRIAL: NCT03761680
Title: MEDPass Trial: MEDPass Versus Conventional Administration of Oral Nutritional Supplements: A RCT Comparing Energy and Protein Intake
Brief Title: MEDPass Trial: MedPass Versus Conventional Administration of Oral Nutritional Supplements
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Bern University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3804
Record Dates: First submitted 2018-11-23; First posted 2018-12-03 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Malnutrition
Keywords: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, open-label, clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MEDPass Group (Experimental): Allocation of ONS in the MEDPass mode
  Interventions: Dietary Supplement: MEDPass mode of administration
- Control Group (Active Comparator): Patients receive ONS between meals or at their request as usual
  Interventions: Dietary Supplement: Control Intervention

INTERVENTIONS:
Dietary Supplement: MEDPass mode of administration — Allocation of 50 ml of ONS four times per day distributed with the medication rounds
  Arms: MEDPass Group
Dietary Supplement: Control Intervention — Patients receive ONS between meals or at their request as usual
  Arms: Control Group

SUMMARY:
The aim of the randomized-controlled, single-center MEDPass trial is to assess the effects of MEDPass versus conventional administration of oral nutritional supplements (ONS) on energy and protein intake in medical and geriatric inpatients.

DETAILED DESCRIPTION:
Disease related malnutrition (DRM) in hospitalized patients is a common problem.The oral nutritional support with ONS is one of the first and most common treatment approach in the patients at nutritional risk. Treatment with ONS may reduce mortality and complications in hospitalized patients.

There are no standards on the type of administration of ONS in terms of timing throughout the day leading to individual approaches. ONS are conventionally served as snacks by nurses, nursing aids or gastronomy personnel between the main meals. The MEDPass-mode offers a different approach by serving ONS together with the medication, three or four times per day, in unusually small portions. Preliminary trials suggest that compliance and cost effectiveness may be improved with the MEDPass-mode.

Enhancing compliance to ONS may not consequently lead to improved total energy and protein intake throughout the day. There has never been a large trial in which total energy- and protein intake of the subjects was studied consequently and systematically throughout the hospitalization. Therefore, this trial will bridge this gap by studying total energy- and protein intake as primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Nutritional risk screening (NRS-2002) total score ≥3 points according to routine screening at admission within 72 hours
* Expected hospital LOS ≥3 days after screening (as estimated by the treating physician)
* Patient qualifies for ONS and approves prescription
* Age >18 years
* Willingness and ability to provide informed consent

Exclusion Criteria:

* Initially admitted to critical care unit
* Immediate post-operative phase (<7 days post-surgery)
* Dysphagia with the inability to swallow liquids
* Supplemental enteral and/or parenteral nutrition
* Admitted with, or scheduled for, total parenteral nutrition or tube feeding
* Mini Mental State examination < 16 points
* hospitalized due to anorexia nervosa
* hospitalized due to acute pancreatitis
* hospitalized due to acute liver failure
* cystic fibrosis
* patients after gastric bypass surgery
* patients with short bowel syndrome
* terminal condition (end of life situation)
* poor skills in German language (study language)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2018-11-22 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Average intake of energy / day (kcal, % of calculated daily requirement) | throughout the hospitalization: min. 3 to max. 30 days

SECONDARY OUTCOMES:
Average intake of protein /day (g, % of calculated daily requirement) | throughout the hospitalization: min. 3 to max. 30 days
Average intake of ONS / day (ml) | throughout the hospitalisation: min. 3 to max. 30 days
Development of hand grip strength (kg) | throughout the hospitalisation: min. 3 to max. 30 days
  Monitored at day 1, day 8, day 15, 22 and 29 or at discharge if at least 5 days after the last measurement have past.
  Evaluated with the JAMAR® Hydraulic Hand Dynamometer (Patterson Medical, Warrenville, IL, USA).
  If possible, measurements are conducted on the dominant hand, three times with a break of at least 30 seconds between the measurements.
  The highest value is noted. Accuracy: 0.5 kg. Range: 0.0 - 90.0 kg
Changes in body weight (kg) | throughout the hospitalisation: min. 3 to max. 30 days
  Monitored at day 1, day 8, day 15, 22 and 29 or at discharge if at least 5 days after the last measurement have past.
  Accuracy: 0.1 kg.
Development of appetite visual analogue scale (VAS)-score (cm) | throughout the hospitalisation: min. 3 to max. 30 days
  Monitored at day 1, day 8, day 15, 22 and 29 or at discharge if at least 5 days after the last measurement have past.
  The present day is the focus of the assessment. On the front of the scale which is visible to the patient, only smileys are shown.
  The scale on the back ranges from 0-10 cm to objectify the measurement with 10 cm being the most desirable.
  Accuracy:0.1 cm.
Development of nausea visual analogue scale (VAS)-score (cm) | throughout the hospitalisation: min. 3 to max. 30 days
  Monitored at day 1, day 8, day 15, 22 and 29 or at discharge if at least 5 days after the last measurement have past.
  The present day is the focus of the assessment. On the front of the scale which is visible to the patient, only smileys are shown.
  The scale on the back ranges from 0-10 cm to objectify the measurement with 10 cm being the most desirable.
  Accuracy: 0.1 cm.
Hospital length of stay (LOS) | hospitalization, max. 30 days
Mortality | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Zeno Stanga, Prof.Dr.med., Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Inselspital, Berne, Facility Tiefenau, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kurmann S, Reber E, Schonenberger KA, Schuetz P, Uhlmann K, Vasiloglou MF, Schoenenberger AW, Bertschi D, Sterchi AB, Stanga Z. MEDPass versus conventional administration of oral nutritional supplements - A randomized controlled trial comparing coverage of energy and protein requirements. Clin Nutr. 2023 Feb;42(2):108-115. doi: 10.1016/j.clnu.2022.11.015. Epub 2022 Dec 5. PMID 36525797
- [Derived] Kurmann S, Reber E, Vasiloglou MF, Schuetz P, Schoenenberger AW, Uhlmann K, Sterchi AB, Stanga Z. Energy and protein intake in medical and geriatric inpatients with MEDPass versus conventional administration of oral nutritional supplements: study protocol for the randomized controlled MEDPass Trial. Trials. 2021 Mar 16;22(1):210. doi: 10.1186/s13063-021-05145-4. PMID 33726841